CLINICAL TRIAL: NCT01596101
Title: Role of Circadian Rhythm of Melatonin on Sleep-related Disturbances Postburn
Brief Title: Circadian Rhythm of Melatonin in Burns
Acronym: Sleep4
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Director, Nutrition Services, Shriners Hospitals for Children
Other Study IDs: 08-07-21-03
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Sleep; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- acute burns
- rehab patients

SUMMARY:
Evaluate markers and postulated effectors of the endogenous circadian pacemaker in children admitted to the burn intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* 5-18 years old

Exclusion Criteria:

* anoxic brain injury
* preexisting neurological disorder
* pre-existing sleep disorder
* no informed consent or HIPAA release

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pediatric burn patients
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2009-04; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
sleep status | 48hrs
  actigraphy, polysomnography

SECONDARY OUTCOMES:
urinary melatonin | every 2 hours for 48 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospital for Children, Cincinnati, Ohio, United States